CLINICAL TRIAL: NCT00424138
Title: [18F]FDG-PET/CT as a Predictive Marker of Tumor Response and Patient Outcome: Prospective Validation in Non-Small Cell Lung Cancer
Brief Title: FDG-PET/CT Scans in Patients With Stage IIIB or Stage IV NSCLC Undergoing Chemotherapy
Acronym: ACRIN6678
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment obstacles; data to be combined with other resources for analysis
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000527084; ACRIN-6678 (Other: ACRIN Foundation); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A - 3 FDG-PET/CT Scans (Experimental): Two FDG-PET/CT scans prior to 1st cycle of chemotherapy, plus 2 optional volumetric CT scans. One FDG-PET/CT after 1st cycle of chemotherapy, plus 1 optional volumetric CT scan.
  Interventions: Radiation: FDG
- Group B - 2 FDG-PET/CT + 1 Optional (Experimental): One FDG-PET/CT prior to 1st cycle of chemotherapy; 1 FDG-PET/CT after the 1st cycle of chemotherapy; 1 optional FDG-PET/CT after the 2nd cycle of chemotherapy. All three with optional volumetric CT scans.
  Interventions: Radiation: FDG
- Group C - Test-Retest (Experimental): Test-retest sequence for FDG-PET/CT; two scans with optional volumetric CT to be completed prior to 1st cycle of chemotherapy.
  Interventions: Radiation: FDG

INTERVENTIONS:
Radiation: FDG
  Other Names: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as fludeoxyglucose F 18 (^18FDG) positron emission tomography (PET)/CT scans, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying ^18FDG PET/CT scans to see how well they predict response in patients undergoing chemotherapy for stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a metabolic response, defined as a 25% decrease in peak tumor standardized uptake value (SUV) after the first course of chemotherapy, provides early prediction of treatment outcome (tumor response and patient survival) in patients with stage IIIB or IV non-small cell lung cancer undergoing platinum-based chemotherapy.
* Determine the test-retest reproducibility of quantitative assessment of tumor fludeoxyglucose F 18 (^18FDG) uptake in these patients.
* Determine the time course of treatment-induced changes in tumor ^18FDG uptake in these patients.
* Determine, in an exploratory analysis, changes in tumor volume during chemotherapy by multislice CT scanning in these patients.

OUTLINE: This is a prospective, multicenter study. Patients are assigned to 1 of 3 groups.

* Group I: Patients undergo fludeoxyglucose F 18 (^18FDG) positron emission tomography (PET)/CT scanning twice and 1-2 volumetric CT scanning (1-7 days apart) before starting treatment with platinum-based chemotherapy. Patients undergo additional ^18FDG PET/CT scan and a volumetric CT scan once between the first and second course of chemotherapy.
* Group II: Patients undergo ^18FDG PET/CT scan and volumetric CT scanning once before starting treatment with platinum-based chemotherapy. Patients undergo additional ^18FDG PET/CT scan and volumetric CT scanning once between the first and second course of chemotherapy, and may undergo once between the second and third course of chemotherapy.
* Group III: Patients undergo ^18FDG PET/CT scanning twice (up to 1 week apart) before starting any treatment.

In groups I and II, patients also undergo standard follow-up CT scanning every 6 weeks (i.e., every other chemotherapy course) for up to 18 weeks.

After completion of chemotherapy, patients are followed every 3 months for up to 1 year.

Biomarker

* Imaging: See
* provided by American College of Radiology Network.

PROJECTED ACCRUAL: A total of 285 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Newly diagnosed stage IIIB (with malignant pleural effusion) or stage IV disease (Group I and II), or newly diagnosed stage IIIA, IIIB, or IV (Group III) determined by all of the following:

    * CT scan or MRI of the chest and upper abdomen (including liver and adrenal glands) within the past 4 weeks
    * History/physical examination within the past 6 weeks
    * CT scan or MRI of the brain within the past 4 weeks, if there is headache, mental/physical impairment, or other signs or symptoms suggesting brain metastases within the past 2 months
  * No small cell carcinoma
  * No pure bronchioloalveolar carcinoma
* Patients with recurrent or metastatic disease are eligible provided they meet 1 of the following criteria:

  * Received surgery or radiotherapy for treatment of the primary tumor and locoregional disease ≥ 3 months prior to study entry AND have a measurable lesion in the chest
  * Received chemotherapy in the adjuvant setting or as part of combined modality therapy for locoregional disease ≥ 3 months prior to recurrent or metastatic disease diagnosis AND have a measurable lesion in the chest
* Measurable disease, defined as at least 1 measurable primary tumor or other intrathoracic/supraclavicular lesion ≥ 2 cm
* Scheduled to be treated with a platinum-based dual-agent chemotherapy regimen administered at 3-week intervals with or without bevacizumab or cetuximab (Group I and II)
* Scheduled to be treated with standard chemotherapy in the current protocol, other standard chemotherapy, experimental chemotherapy, or other treatment including no treatment (Group III)
* No symptomatic brain metastases (Groups I and II only)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2 (Groups I and II only)

  * Group III may include potential participants regardless of ECOG performance status score
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to tolerate positron emission tomography (PET)/CT scanning
* No contraindication to chemotherapy and PET/CT scanning, as demonstrated by laboratory testing
* No poorly controlled diabetes (i.e., fasting glucose level > 150 mg/dL) despite attempts to improve glucose control by fasting duration and adjustment of medications
* No prior malignancy other than basal cell or squamous cell carcinoma of the skin, carcinoma in situ, or other cancer from which the patient has been disease free for ≥ 3 years (Groups I and II)

  * Prior malignancy is not an exclusion factor for Group III
* No clinical or radiographic signs of post-obstructive pneumonia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior thoracic radiotherapy, lung surgery, or chemotherapy
* Prior chemotherapy in the adjuvant setting or as part of a combined modality regimen for locoregional disease that was given ≥ 3 months prior to diagnosis of recurrent or metastatic disease allowed
* No planned treatment with any targeted biologic therapy including gefitinib or erlotinib hydrochloride (Group I and II)
* No concurrent chemoradiotherapy
* No concurrent bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-03-30 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
Prediction of 1-year overall survival as measured by monitoring changes in tumor metabolic response during the first course of chemotherapy | One year

SECONDARY OUTCOMES:
Correlation of metabolic response after the first course of chemotherapy with subsequent best tumor response as measured by RECIST criteria | 1st Course Chemotherapy
Correlation of metabolic response after the first course of chemotherapy with progression-free survival | 1st Course of Chemotherapy
Predictive value of fludeoxyglucose F 18 positron emission tomography (FDG-PET) for 1-year overall survival after the first and second course of chemotherapy | One year
Test-retest reproducibility of standardized uptake values (SUV) as measured by FDG-PET/CT scans | Within 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Weber, MD, Study Chair — Jonsson Comprehensive Cancer Center; Denise R. Aberle, MD, Study Chair — Jonsson Comprehensive Cancer Center; Barry A. Siegel, MD, Study Chair — Washington University Siteman Cancer Center; Anthony F. Shields, MD, PhD, Study Chair — Barbara Ann Karmanos Cancer Institute; Karen Rickard, Study Chair — City of Hope Comprehensive Cancer Center; Ramaswamy Govindan, MD, Study Chair — Washington University Siteman Cancer Center; Steven M. Dubinett, MD, Study Chair — Jonsson Comprehensive Cancer Center; Joel Karp, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
See ACRIN data sharing policy:
  https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- See also: National Cancer Institute's clinical trials database — https://clinicaltrials.gov/ct2/show/NCT00424138